CLINICAL TRIAL: NCT02386293
Title: Effectiveness of Avapro in the Treatment of Salt Sensitivity in Both Normotensive and Untreated Hypertensive Obese African Americans: A Randomized Double Blind Placebo Controlled Trial
Brief Title: Effectiveness of Avapro in Obese Normotensive/Hypertensive African Americans
Acronym: Avapro3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Gregory Harshfield, Director, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 611881
Record Dates: First submitted 2015-03-03; First posted 2015-03-11 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Hypertension; Obesity; Stress, Psychological; Blood Pressure
MeSH Terms: conditions — Hypertension; Obesity; Stress, Psychological | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Sugar pill identical to Avapro provided for 7 day prescription
  Interventions: Other: Placebo
- Irbesartan (Active Comparator): 150 mg of Avapro once daily for 7 days.
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: Irbesartan — Double blind placebo controlled cross over trial to determine effectiveness of an angiotensin receptor blocker in obese hypertensive African American patients.
  Other Names: Avapro
  Arms: Irbesartan
Other: Placebo — Sugar pill made to look identical to irbesartan intervention.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that hypertension increases the anti-natriuretic effects of an angiotensin receptor antagonist during mental stress in overweight/obese African-American's who retain sodium during mental stress.

DETAILED DESCRIPTION:
Using a crossover design, we will compare the effects of a placebo to an angiotensin II receptor antagonist on the urinary sodium excretion response in obese normotensive subjects and untreated hypertensive African-Americans subjects. We expect that the urinary sodium excretion response to angiotensin II receptor antagonist therapy will be less in the overweight/obese hypertensive subjects compared to the overweight/obese normotensive subjects. This study will also employ a double blind placebo controlled cross-over drug study. Half of the subjects will be normotensive and half drug naïve hypertensive. The normotensive subjects will be identified as described above for Studies 1 and 2. The hypertensive subjects will be identified by Dr. White or his team in the hypertension clinic. These patients will be restricted to those not currently on anti-hypertensive therapy.

This study will involve a screening visit, two first dose visits and two testing weeks over an approximate 5 week period (this includes a one week "washout" period).

Each testing week will have a 3 day salt-controlled diet prior to testing and an approximate 3-hour testing period on Day 4. The 3-hour testing period will include 10 minutes of a baseline rest, 45 minutes of mild stress (competitive video game), and 45 minutes of a recovery rest. A total of 4 blood and 4 urine samples will be collected during the 3-hour period. Each blood draw will consist of about 7 teaspoons for a total of 28 teaspoons per week. If female, a pregnancy test will be performed at the beginning of each testing visit (screening, first dose-1, test day-1, first dose -2 and test day-2) to confirm that they are not pregnant. The week before testing, the subject will come to the Georgia Prevention Institute or Children's Research Unit for the First Dose Visit and meet with one of the study physicians who will give me instructions on how to take Avapro. This appointment will last about 2 ½ hours. They will take their first dose of Avapro or the placebo and will be monitored for the next 2 hours. If female subject, they will provide a urine sample for a pregnancy test to make sure they are not pregnant before they are given the first dose of the study medication. During this time, their blood pressure will be taken every 15 minutes.

During the screening and testing, each subject will be asked to take the MoCA (the Montreal Cognitive Assessment) test in order to measure cognitive thinking after stress. It is a brief 30-question test which takes around 10 minutes to complete. It measures different types of cognitive abilities, including orientation (the approximate position of something/someone), short-term memory (remember information for a short period of time), executive function (planning and problem solving), language abilities (assign appropriate names to appropriate items), and visuospatial ability (determine distance from one object to another). Each question is awarded a particular number of points depending on the accuracy of the answers given. We will be looking to see if the total number of points earned changes in response before and after stress. During the screening visit, they subject will take the MoCA test which will take approximately 10 minutes. Someone from the research team will instruct the subject as to what to do for each question and they will answer each one to the best of their ability.

On testing day, a nurse/phlebotomist will insert a small needle attached to a plastic tube called a catheter into a vein in the hand or arm. This procedure will allow the nurse/phlebotomist to collect the 4 blood samples over the 3-hour testing period. The needle stick may cause some temporary pain and may result in a black and blue mark. A device that automatically takes blood pressure will then be put on the opposite arm. The subject will also be given water to sip on during the duration of testing. Before testing begins, the subject be instructed to take their last dose of medication. During the first 10 minute baseline rest period, they will relax in a reclining chair. They can listen to music, read a book or magazine or watch movies to pass the time. Blood pressure will be taken before and after this 10 minute rest period. Once the baseline rest period is over, a blood and urine sample will be collected.

During the stress period, the subject will play a video game against another subject for 45 minutes. Blood pressure will continue to be measured every 10 minutes. They will also continue to sip on water during this time. At the end of the game, another blood and urine sample will be collected.

The subject will then be asked to complete the MoCA test a second time. It will be the same questions that was asked during the screening visit. A research team member will instruct the subject again as to how to answer each question and they will answer them to the best of their ability.

The last 45 minute recovery period of relaxation will be the same as the first (reading, listening to music or watching movies). Blood pressure will continue to be taken every 10 minutes. Once the 45 minutes has ended the last blood and urine sample will be collected and the testing day will have been completed. They will repeat this whole process a second time.

During test day one or test day two, each subject will have a Dual Energy X-ray Absorptiometer (DEXA) scan and a Peripheral Quantitative Computer Tomography (pQCT) scan performed on them The DEXA is to assess bone mineral density (BMD), body fat percentage and lean tissue. The pQCT will assess bone strength at the radius and tibia. For The DEXA, the subject will remove any items that may contain metal - including jewelry, belts, shoes and piercings. A gown will be provided if needed. The subject will lie on a table for approximately 6 minutes, while the table rotates and a mechanical arm moves above the subject body measuring for the BMI. For the pQCT, the subject will be seated and position their forearm into the pQCT device and remain still for 3-5 minutes. They will then place their lower leg into the same device for another 3-5 minutes to be scanned. If the subject is female, a pregnancy test will be performed before any testing begins for each testing visit in order to confirm the subject is not pregnant.

Bone and Body Composition Measurements

Dual-energy X-ray absorptiometry will be performed at baseline and posttest to assess total body composition. The body composition variables of interest will be fat-free soft tissue mass and fat mass.

Peripheral quantitative computed tomography will be performed at baseline visit only to assess bone strength at the radius and tibia. During the scan, the participant must place their forearm or lower leg into the pQCT unit and remain still for three to five minutes (actual scan duration for each).

For the forearm scan, the participant is seated in a chair at the side of the pQCT unit. The participant sits as close as possible to the unit. The shoulder should be close to the front side of the gantry. The armrest of the machine is adjusted to the measured forearm length. The elbow is fixed at the corner of the armrest with the Velcro strap and the distal forearm is fixed with the clamp. The angle between upper arm and forearm should not exceed 90°. The hand lies on the hand rest. The fixation of the arm should prevent movement artifacts but must not hurt. The participant is asked to search for a convenient and natural position to avoid movement or discomfort during the scanning period of 3-5 minutes.

For the lower leg scan, the participant is seated on a chair in front of the pQCT unit. When the machine is at the start position, the participant's lower leg is moved through the gantry and the foot is rested on the foot holder. With the foot holder positioned all the way to the front of the pQCT unit, the lower leg is centered and fixed into the concentric acrylic cylinder (diameter 18 cm), which is located at the gantry opening. The foot is now fixed with the Velcro strap to the foot holder. Before the scan, the participant is asked to find a convenient and natural position to reduce movement artifacts during the 3-5 minute scan.

Radial and tibial measurements will be taken at the 4% and 20% sites for bone outcomes, proximal to the articular surface of the distal end of the tibia and radius. The 4% and 20% sites represent areas high in trabecular and cortical bone, respectively. Each scan will be acquired with a 0.4 mm voxel size and a slice thickness of 2.4 mm. The anatomic reference line (for determination of the distal end of the radius or tibia) will be identified by acquisition of a 30 mm planar scout view of the joint line and automatically set by the software at 4% or 20% sites. Image processing and calculation of the bone measures will be determined using the Stratec software (version 6.02 d).

At the trabecular sites of the radius and tibia, total volumetric bone mineral density (vBMD, mg/cm3) and total cross-sectional area (CSA, mm2) will be measured to calculate bone strength index (BSI; mg2/mm4, Equation 1), an estimate of bone's ability to withstand compressional strains. At the cortical bone sites of the radius and tibia, cortical vBMD (mg/cm3), cortical CSA (mm2), and cortical thickness (mm) will be measured to calculate the strength-strain index (SSI, mm3), which reflects torsional bone strength. The SSI is calculated as the integrated product of the section modulus and the density of cortical bone (Equation 2). Section modulus is calculated as (a x d2)/dmax, where a is the CSA of a voxel, d is the distance of the voxel from the center of gravity, and dmax is the maximum distance of one voxel to the center of gravity. The ratio of cortical vBMD and normal physiological density (ND = 1200 mg/cm3) provides an estimate of the modulus of elasticity.

ELIGIBILITY:
Inclusion Criteria:

* of good general health
* not on any prescription medications
* between the ages of 18 and 50
* not pregnant

Exclusion Criteria:

* not African-American
* pregnant
* taking medications that will affect my blood pressure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Urinary sodium excretion rate | 2 hours
  primary variable of interest is the difference in stress induced changes in sodium excretion between placebo and treatment conditions in obese normotensives versus non-obese hypertensives.

SECONDARY OUTCOMES:
Hemodynamics | 2 hours
  measures of change in systolic blood pressure compared to changes in sodium excretion in treatment versus placebo in obese normotensives versus non-obese hypertensives.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Harshfield, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Dissemination will be carried out in a variety of ways that will be accessible to other scientists studying psychosocial stress, hypertension, and the control of fluid-electrolyte balance and blood pressure. These include publications made available through PubMed-cited journals and presentations at scientific meetings and various organizations.
Supporting Information: Study Protocol